CLINICAL TRIAL: NCT05147454
Title: Assessing Somatosensory System Damage in Trigeminal Neuralgia and Persistent Idiopathic Facial Pain Through Neuroimaging and Quantitative Sensory Testing
Brief Title: MRI & QST Analysis in Trigeminal Neuralgia and Persistent Idiopathic Facial Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Walton Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG447-21
Record Dates: First submitted 2021-10-18; First posted 2021-12-07 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Facial Pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trigeminal Neuralgia: Patients with a definite diagnosis of Classical or Idiopathic Trigeminal Neuralgia
  Interventions: Other: Quantitative Sensory Testing
- Persistent Idiopathic Facial Pain: Patients with a definite diagnosis of Persistent Idiopathic Facial Pain
  Interventions: Other: Quantitative Sensory Testing

INTERVENTIONS:
Other: Quantitative Sensory Testing — Non-invasive assessment of Sensory Profile

SUMMARY:
Patients with a definite diagnosis of classical TGN and PIFP will undergo a structured clinical questionnaire and a trigeminal sensory profile using the quantitative sensory testing. Clinical measures and sensory profiles will be correlated with MRI measures.

DETAILED DESCRIPTION:
Patients with a definite diagnosis of classical TGN and PIFP (according to the 2020 ICOP Classification) will undergo a structured clinical questionnaire and a trigeminal sensory profile using the quantitative sensory testing. Clinical measures and sensory profiles will be correlated with the presence and the geometry of neurovascular compression at MRI. Moreover quantitative structural neuroimaging analysis, such as trigeminal root volume, will be performed in each patient and correlated with clinical and QST data.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of Classical or Idiopathic Trigeminal Neuralgia or Persistent Idiopathic Facial Pain according to the latest ICOP 2020 Criteria
* Naive to any surgical procedures

Exclusion Criteria:

* Any major chronic painful or other neurological disease
* Diagnosis of Secondary Trigeminal Neuralgia
* Diagnosis of other facial pain syndromes
* Cognitive disturbances

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients attending The Walton Centre Clinics
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-07-17 (Estimated); Study Completion 2024-07-17 (Estimated)

PRIMARY OUTCOMES:
Sensory Profile | Baseline, at the time of visit
  Sensory Profile as assessed by Quantitative Sensory Testing

SECONDARY OUTCOMES:
Presence of Neurovascular Compression | Baseline, at the time of visit
  Presence of Neurovascular Compression defined as absence of any liquor cleft between the trigeminal root and the offending vessel, on dedicated Trigeminal MRI
Trigeminal Root Volume | Baseline, at the time of visit
  Trigeminal Root Volume as assessed by specific neuroimaging Software (MIPAV)
Geometry of Neurovascular Compression | Baseline, at the time of visit
  Measurement of the polar coordinates beetween the trigeminal root and the offending vessel as assessed by specific neuroimaging Software (MIPAV)

CONTACTS AND LOCATIONS:
Locations (1):
- The Walton Centre NHS Foundation Trust, Liverpool, United Kingdom